CLINICAL TRIAL: NCT06786000
Title: Neurophysiological and Behavioral Effects of Combining Transcranial Direct Current Stimulation (tDCS) and Modified-Constraint Induced Movement Therapy (mCIMT) on Upper Limb Function Recovery in Patients with Stroke
Brief Title: Neurophysiological and Behavioral Effects of Combining Transcranial Direct Current Stimulation (tDCS) and Modified-Constraint Induced Movement Therapy (mCIMT)
Acronym: tDCS and mCIMT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Collaborators: King Saud Medical City (Other Government); King Fahad Medical City (Other Government)
Responsible Party: Principal Investigator, Dr. Alaa Albishi, Associate Professor, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-23-7495
Record Dates: First submitted 2025-01-02; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Stroke; Hemiparesis of the Upper Limb Following Stroke; Stroke Rehabilitatiom
Keywords: stroke; ischemic stroke; hemorrhagic stroke; tDCS; mCIMT; hemiparesis; neural activation; primary motor cortex; NIBS; non invasive brain stimulation; trans direct current stimulation; modified constraint induced movement therapy
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke; Paresis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Anodal tDCS combined with mCIMT (Experimental): 20 minutes of anodal tDCS followed by 1 hour of the mCIMT program
  Interventions: Device: Anodal tDCS combined with mCIMT
- Cathodal tDCS combined with mCIMT (Experimental): 20 minutes of cathodal tDCS followed by 1 hour of the mCIMT program
  Interventions: Device: Cathodal tDCS combined with mCIMT
- Bihemispheric tDCS combined with mCIMT (Experimental): 20 minutes of bihemispheric tDCS followed by 1 hour of the mCIMT program
  Interventions: Device: Bihemispheric tDCS combined with mCIMT
- Sham tDCS combined with mCIMT (Sham Comparator): 20 minutes of anodal tDCS (after 30 seconds of stimulation, the stimulator will switch off) followed by 1 hour of the mCIMT program
  Interventions: Device: Sham tDCS combined with mCIMT

INTERVENTIONS:
Device: Anodal tDCS combined with mCIMT — 20 minutes of anodal tDCS followed by 1 hour of the mCIMT program. The anodal electrode will be placed over the ipsilesional M1 (primary motor cortex, C3 or C4 according to EEG 10/20 system), and the cathodal electrode over the contralateral supraorbital area (Fp1 or Fp2) ). Leading to subthreshold depolarization to promote cortical excitation. And twelve different oriented tasks will be used during the 1-hour training period.
  Arms: Anodal tDCS combined with mCIMT
Device: Cathodal tDCS combined with mCIMT — 20 minutes of cathodal tDCS followed by 1 hour of the mCIMT program. the cathodal electrode will be placed over the contralesional M1, and the anodal electrode over the contralateral supraorbital area (Fp1 or Fp2). leading to subthreshold polarization to promote cortical inhibition. And twelve different oriented tasks will be used during the 1-hour training period.
  Arms: Cathodal tDCS combined with mCIMT
Device: Bihemispheric tDCS combined with mCIMT — 20 minutes of Bihemispheric tDCS followed by 1 hour of the mCIMT program. the cathodal electrode will be placed over the primary motor cortex (M1) of the contralesional hemisphere and the anodal electrode will be placed above the ipsilateral M1 position (C3 or C4 positions, according to the 10/20 EEG system). And twelve different oriented tasks will be used during the 1-hour training period.
  Arms: Bihemispheric tDCS combined with mCIMT
Device: Sham tDCS combined with mCIMT — 20 minutes of sham tDCS followed by 1 hour of the mCIMT program. the same stimulation place and parameters will be used as in the anodal group. However, after 30 seconds of stimulation, the stimulator will switch off. This provides the participants with the experience of the initial itchy sensation that occurs during tDCS, which is required for efficient masking. And twelve different oriented tasks will be used during the 1-hour training period.
  Arms: Sham tDCS combined with mCIMT

SUMMARY:
This clinical trial aims to evaluate the effect of different types of tDCS modulation with mCIMT in improving affected upper-limb motor function for stroke patients. The main question it seeks to answer:

Which type of tDCS (bi-hemispheric, anodal, or cathodal) combined with the mCIMT program leads to greater improvement in affected upper-limb function in patients with stroke? Researchers will compare these three types of tDCS to a sham tDCS. To see which kind of tDCS protocol combined with the mCIMT program will be more effective in improving affected upper-limb function for stroke patients.

Participants will:

1. Participants will receive 12 sessions of mCIMT combined with tDCS or mCIMT alone.
2. Visit the clinic three times a week for four weeks.
3. Participants will do fMRI and TMS before and after the program and three times of assessment before and after two weeks after the program.

DETAILED DESCRIPTION:
Background: After a stroke, intense motor rehabilitation is required to facilitate motor recovery. In specific, combining tDCS with neurorehabilitation interventions boosts the responses of the brain to the interventions and maximizes the effects of rehabilitation to improve upper limb recovery post-stroke. Objectives: To evaluate the effect of different modes of tDCS modulation with mCIMT in improving affected upper-limb motor recovery for patients with stroke. Method: a randomizing control trial design, after performing a baseline assessment, the participants will be randomly assigned to one of the four groups: the anodal tDCS +mCIMT group, the cathodal tDCS +mCIMT group, the bihemispheric tDCS +mCIMT group, and the mCIMT alone group. Inclusion Criteria, adult participants clinically diagnosed and confirmed by imaging of ischemic or hemorrhagic cerebrovascular accident, participant's age older than 18 years, Stroke onset more than 3 months with unilateral motor deficits, Adequate cognitive function is required to follow instructions. The Arabic version of the Mini-Mental State Examination (MMSE) should be ≥24, 10° of active extension to the metacarpophalangeal and interphalangeal joints and 20° at the wrist, and not participating in other clinical, or research studies at the same time. Exclusion Criteria, Severe muscle spasticity at the affected limb at all joints (the Modified Ashworth Scale scores > 3), Contraindications to NIBS, unilateral neglect, Other neurologic or orthopedic conditions that may affect hand function, and unstable medical conditions. The total intervention period will be performed 3 times a week for 4 weeks. Each participant will undergo motor impairment and physiological assessments at baseline, during and after the intervention. Functional outcome measures: Fugl-Meyer Assessment Scale - upper extremity (FMA-UE), Wolf Motor Function Test (WMFT), Nine-Hole Peg Test (NHPT), Arabic version of Stroke Impact Scale (SIS-16), and Stroke-Specific Measure of Adherence to Home-based Exercises (SS-MAHE). Physiological outcome measures: Cortical Excitability Assessment will be measured by Transcranial Magnetic Stimulation (TMS) with electromyographic (EMG) and functional magnetic resonance imaging (fMRI).

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants clinically diagnosed and confirmed by imaging of ischemic or hemorrhagic cerebrovascular accident (Dahl et al., 2008; Jin et al., 2019).
2. Participant's age older than 18 years (Baltar et al., 2020).
3. Stroke onset more than 3 months with unilateral motor deficits (Lin et al., 2010).
4. Adequate cognitive function is required to follow instructions. The Arabic version of the Mini Mental State Examination (MMSE) should be ≥24 (Kim, 2021).
5. 10° of active extension to the metacarpophalangeal and interphalangeal joints and 20° at wrist will be assessed by manual goniometer (Dahl et al., 2008).
6. Fugl-Meyer assessment (FMA) scores between 19 and 58, indicating moderate to mild impairments.
7. Not participating in other clinical, or research studies at the same time.

Exclusion Criteria:

1. Severe muscle spasticity at the affected limb at all joints (the Modified Ashworth Scale scores > 3) (Baltar et al., 2020).
2. Contraindications to NIBS (Bornheim et al., 2019).
3. Unilateral neglect (Dahl et al., 2008)
4. Other neurologic or orthopedic conditions that may affect hand function.
5. Unstable medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-04-11 (Actual); Primary Completion 2025-04-11 (Estimated); Study Completion 2025-04-11 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment Scale - upper extremity (FMA-UE) | at baseline, and after 2 weeks, and after intervention (4 weeks).
  The upper extremity domain of FMA consists of 33 items (reflex activity, volitional movement within synergies, volitional movement mixing synergies, volitional movement with little or no synergy, wrist, hand, coordination/ speed). On a 3-point ordinal scale, 0 = cannot perform, 1 = performs partially, and 2 = performs fully. The upper extremity domain has a total score of 66. A higher score indicated better performance of the affected side.
Wolf Motor Function Test (WMFT) | at baseline, and after 2 weeks, and after intervention ( 4 weeks).
  It is used to assess upper-limb performance through timed and functional tasks (Wolf et al., 2001). The WMFT is preferred to frequently used upper limb performance tests since it assesses a wide range of functional activities (from simple to complex) and investigates both performance time and movement quality (Morris et al., 2001). The modified WMFT consists of 17 items, 2 of which are strength measurements, and the remaining 15 items are functional tasks that gradually progress from simple movements in the proximal joint to complex movements in the distal joint. Each of the 15 tasks is timed to completion, up to a maximum of 120 seconds (Wolf et al., 2001). The items are scored on a 6-point scale ranging from 0 (does not attempt with the upper limb being tested) to 5 (uses the limb being tested, movement appears normal) (Wolf et al., 2005). A lower score indicates a lower functional level (Wolf et al., 2005).
Nine-Hole Peg Test (NHPT) | at baseline, and after 2 weeks, and after intervention ( 4 weeks).
  The Nine-Hole Peg Test (NHPT) is one of the most commonly used performance tests for measuring hand function and manual dexterity in stroke patients (Chen et al., 2009; Mathiowetz et al., 1985). The NHPT consists of a container with nine pegs and a pegboard with nine holes. The board will be placed at the midline of the patient, with the container containing the pegs on the side of the hand being evaluated. The NHPT requires the patient to pick up the pegs from the container with the affected upper limb, transfer and insert them into the holes of the pegboard until it is full, and then return them to the container. Patients will be instructed to complete the test as quickly and accurately as possible (Sommerfeld et al., 2004). The score will be based on the time it takes to complete the test activity, which will be recorded in seconds. The stopwatch should be started when the patient touches the first peg until the last peg is put in the container (Oxford Grice et al., 2003).
Cortical Excitability Assessment | at baseline and after intervention ( 4 weeks).
  The Transcranial Magnetic Stimulation (TMS) will be used to assess the corticospinal excitability through the measurement of the TMS-elicited motor evoked potential (MEP) in both the lesioned and the nonlesioned motor cortices (Wassermann et al., 2008). Online monitoring of the electromyographic (EMG) activity in response to TMS will be performed, MEPs will be recorded from the left and the right first interosseous (FDI) muscles
Functional magnetic resonance imaging (fMRI) | at baseline and after intervention ( 4 weeks).
  Functional magnetic resonance imaging (fMRI) is a type of magnetic resonance imaging (MRI) that measures brain activity and connectivity. During an fMRI scan, a block design will be used. Each scan will take 6 minutes and be split into six blocks in the following order, with a rest of 30 seconds between each of the 15 contractions that last 2 seconds each and 30 seconds of rest in between (Wen et al., 2014). In each task, participants will be asked to grip a rubber ball at a target pressure of 30% of their maximum voluntary contraction using their affected hand (Cheng et al., 2021; Ismail et al., 2014). Visual feedback will be provided for the patients to guide the movement (Könönen et al., 2012).
Wolf Motor Function Test (WMFT) | at baseline and after intervention ( 4 weeks).
  It is used to assess upper-limb performance through timed and functional tasks (Wolf et al., 2001). The WMFT is preferred to frequently used upper limb performance tests since it assesses a wide range of functional activities (from simple to complex) and investigates both performance time and movement quality (Morris et al., 2001). The modified WMFT consists of 17 items, 2 of which are strength measurements, and the remaining 15 items are functional tasks that gradually progress from simple movements in the proximal joint to complex movements in the distal joint. Each of the 15 tasks is timed to completion, up to a maximum of 120 seconds (Wolf et al., 2001). The items are scored on a 6-point scale ranging from 0 (does not attempt with the upper limb being tested) to 5 (uses the limb being tested, movement appears normal) (Wolf et al., 2005). A lower score indicates a lower functional level (Wolf et al., 2005).

SECONDARY OUTCOMES:
Arabic version of Stroke Impact Scale (SIS-16) | at baseline, and after 2 weeks, and after intervention ( 4 weeks).
  Stroke Impact Scale (SIS-16) is a stroke specific, self-reported outcome measure used to assess the impact of stroke on health-related quality of life status related to physical function (P. Duncan et al., 2003). It consists of 16 items, basic and instrumental activities of daily living (7 items), mobility (8 items), and hand function (1 item) on a 5-level Likert scale, 1 = inability to complete the item; 5 = not difficult at all (P. Duncan et al., 2003; P. W. Duncan et al., 2003). Higher scores indicate a better level of health-related quality of life status for stroke patients (P. W. Duncan et al., 2003).
Motor Activity log (MAL) | at baseline, week 1, week 2, week 3 and after intervention ( 4 weeks).
  The MAL consists of two scales; amount of use (AOU), which is the amount the stroke patient uses on the affected limb, and quality of movement (QOM), which is the patient's perceived quality of movement while performing 30 items of daily life (Taub et al., 1993). The items are scored on a 6-point scale ranging from 0 (did not use my weaker arm) to 5 (used my weaker arm as often as before the stroke) for measuring AOU; and to measure QOM, the patient is asked how well the affected limb helped during this activity. Possible scores range from 0 (my weaker arm was not used at all for that activity) to 5 (the ability to use my weaker arm for that activity was as good as before the stroke) (Taub et al., 1993).

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University Medical City, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baltar A, Piscitelli D, Marques D, Shirahige L, Monte-Silva K. Baseline Motor Impairment Predicts Transcranial Direct Current Stimulation Combined with Physical Therapy-Induced Improvement in Individuals with Chronic Stroke. Neural Plast. 2020 Nov 25;2020:8859394. doi: 10.1155/2020/8859394. eCollection 2020. PMID 33299400